CLINICAL TRIAL: NCT02328105
Title: LCI-LUN-ABR-001: A Pilot Study of Carboplatin With Nab-Paclitaxel in Patients With Advanced Non-Small Cell Lung Cancer of Squamous Histology
Brief Title: LCI-LUN-ABR-001: Carbo With Nab-Paclitaxel in Patients With Advanced NSCL Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCI-LUN-ABR-001; 00010224
Record Dates: First submitted 2014-12-17; First posted 2014-12-31 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2021-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carboplatin + Abraxane (Experimental): Carboplatin (AUC = 6; on Day 1) plus Abraxane (nab-paclitaxel; 100 mg/m^2; Days 1, 8, 15) for 6 21-day cycles. Treatment was discontinued if: disease progression, unacceptable toxicity, withdrawn consent, or completion of treatment
  Interventions: Drug: Carboplatin; Drug: Abraxane

INTERVENTIONS:
Drug: Carboplatin — Dosing: AUC = 6; on Day 1
Drug: Abraxane — 100 mg/m^2; Days 1, 8, 15
  Other Names: nab-paclitaxel

SUMMARY:
ABRAXANE, based on results from prior studies, is a promising drug in squamous cell carcinoma of the lung. This study will help to explore the combination of ABRAXANE and carboplatin more thoroughly in the subgroup of patients who had the best response in prior studies as well as determine whether there are any biomarkers which can predict for response.

DETAILED DESCRIPTION:
This is a single arm phase II study for subjects receiving first line therapy for metastatic squamous cell lung cancer. Following informed consent and eligibility check, all subjects will receive therapy with carboplatin and ABRAXANE on an outpatient basis. A total of 50 subjects will be enrolled over an enrollment period of about 24 months. Interim analyses will be conducted after the enrollment of subject 15, subject 30, and subject 45. Tissue biomarkers will be analyzed at baseline; and blood biomarkers will be analyzed at baseline, pre-dose on cycles 3 and 5, and then within 30 days of last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IV non-small cell lung cancer with predominantly squamous histology
* No prior systemic treatment for metastatic disease. Patients who have received prior adjuvant chemotherapy for early-stage lung cancer are eligible if at least 12 months have elapsed between the date of final chemotherapy administration and the date of consent
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or as >10 mm with CT scan, MRI, or calipers by clinical exam
* Biopsy accessible disease
* Patients with previous radiotherapy as definitive therapy for locally advanced non-small cell lung cancer are eligible, as long as the recurrence is outside the original radiation therapy port. Definitive radiation therapy must have been completed >4 weeks prior to the date the informed consent is signed
* Age >18 years
* ECOG performance status less than or equal to 1
* If patient has brain metastasis, the disease must be stable (treated and/or asymptomatic) for at least 4 weeks prior to first dose of study treatment
* Bilirubin < 1.5 mg/dL
* Adequate liver function: AST and ALT <= 2.5x upper limit of normal, alkaline phosphatase <= 2.5x upper limit of normal, unless bone metastasis is present (< 5x upper limit of normal) in the absence of liver metastasis
* Adequate bone marrow function: Platelets >100,000 cells/mm3, Hemoglobin > 9.0g/dL and ANC > 1,500 cells/mm3
* Adequate renal function with creatinine <1.5 mg/dL is recommended
* Females of childbearing potential and sexually active males must use an effective contraception method during treatment and for six months after completing treatment
* Negative serum or urine B-hCG pregnancy test at screening for patients of childbearing potential
* Patients must have < Grade 2 pre-existing peripheral neuropathy (per CTCAE version 4.0)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria

* Received prior systemic therapy for metastatic disease
* Received limited field radiation for palliation <= 2 weeks prior to starting study treatment and/or from whom >= 30% bone marrow was irradiated
* Receiving any other investigational agents
* Known hypersensitivity to either carboplatin or ABRAXANE
* Uncontrolled and current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breast feeding
* Other active malignancies
* Neuropathy greater than or equal to grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-12; Primary Completion 2017-06-15 (Actual); Study Completion 2019-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Mileham, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carboplatin + Abraxane
Started | 11
Completed | 0
Not Completed | 11
Not completed — Death | 6
Not completed — Withdrawal by Subject | 1
Not completed — Still On Study in Follow-Up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Carboplatin + Abraxane
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.09 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
ECOG at Baseline [Count of Participants; unit: Participants] — ECOG Scale of Performance Status, developed by the Eastern Cooperative Oncology Group, where 0 indicates subject is fully active, able to carry on all pre-disease performance without restriction and where 1 indicates subject is restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Participants
    ECOG 0 | 5
    ECOG 1 | 6
Primary Tumor Site - Lung [Count of Participants; unit: Participants] | 11
Tumor Histology - Squamous NSCLC [Count of Participants; unit: Participants] | 11
Stage - IV [Count of Participants; unit: Participants] — Stage of histologically confirmed Non-Small Cell Lung Cancer, per AJCC (American Joint Committee on Cancer) staging criteria
  Participants | 11
Tumor Grade [Count of Participants; unit: Participants] — Grade of tumor per AJCC (American Joint Committee on Cancer) staging criteria
  Participants
    High | 7
    Low | 4
Smoking Status [Count of Participants; unit: Participants]
  Previous Smoker | 7
  Current Smoker | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response
Description: The primary endpoint is a binary variable determined for each patient indicating whether or not they achieved a complete response (CR) or a partial response (PR) as per RECIST 1.1 (where a CR is indicated by disappearance of all target and non target lesions and a PR is indicated by >= 30% decrease in sum of longest diameter of target lesions with baseline as reference). Because overall response is the primary endpoint for this study, best responses of CR or PR must be confirmed by a subsequent radiologic assessment.
Time Frame: Up to a planned 18 weeks
Population: The efficacy population (or evaluable population) is defined as all subjects who have measurable disease present at baseline, have received at least one dose of study therapy, and have had their disease re-evaluated (either clinically or radiographically)
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin + Abraxane
Number analyzed (Participants) | 11
Participants | 4
Statistical Analysis 1: Comparison: Carboplatin + Abraxane; Test type: Superiority — Assuming the true overall response rate is 0.20 under the null hypothesis, then this design will provide 81% power to detect a difference of 0.15 under the alternative hypothesis, assuming a one-sided alpha = 0.09 significance level. A three stage design with n=15, 30 and 45 subjects was determined with the following rejection regions: For n = 15, the rejection region in number of responses (CR or PR) is 0 - 2, for n = 30 it is 3 - 6, and for n = 45 it is 7 - 12; p = 0.161, Fisher Exact — This p-value is only based on partial enrollment of stage 1. As enrollment was halted early, this p-value is descriptive in nature and cannot determine the success/failure of the trial; Response Rate = 0.364, 95% CI 2-sided [0.109 to 0.692] — Confidence interval estimated using the Clopper Pearson method

2. Secondary Outcome: Number of Subjects With Stable Disease or Response
Description: Disease control is calculated for each subject indicating whether or not they achieved an overall response of stable disease or better by RECIST 1.1 (where a CR is indicated by disappearance of all target and non target lesions, a PR is indicated by >= 30% decrease in sum of longest diameter of target lesions with baseline as reference, and SD is neither sufficient shrinkage to qualify for PR nor sufficient growth, >=20%, to indicate progression).
Time Frame: 18 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin + Abraxane
Number analyzed (Participants) | 11
Participants | 9
Statistical Analysis 1: Comparison: Carboplatin + Abraxane; Test type: Other — Estimation only; Disease Control Rate = 0.818, 95% CI 2-sided [0.482 to 0.977] — Confidence interval estimated using the Clopper Pearson method

3. Secondary Outcome: Progression Free Survival
Description: PFS is defined as time from enrollment to time of progression or death. Disease progression (PD) may be determined objectively per RECIST 1.1 (Response Evaluation Criteria in Solid Tumors, where PD is defined as a 20% increase in the sum of longest diameters of target lesions, a measurable increase in non-target lesion, or appearance of new lesions) or subjectively as determined by investigator (with evidence documented in the medical records). If the subject died without documented PD, date of progression will be date of death. For surviving subjects who did not have documented PD, PFS was censored at last radiologic assessment. For subjects who received subsequent anti-cancer therapy prior to documented PD, PFS was censored at last radiologic assessment prior to commencement of subsequent therapy. Subjects who experienced a PFS event following an interval equal to two or more scheduled radiologic assessments were censored at last assessment prior to first missed assessment.
Time Frame: From date of treatment start to date of progression/death, or censored as described above; assessed for approximately 3 years
Population: Efficacy analyses were conducted on the population of subjects who began Carboplatin + Abraxane treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin + Abraxane
Number analyzed (Participants) | 11
months | 7.3 [2.2 to 13]
Statistical Analysis 1: Comparison: Carboplatin + Abraxane; Test type: Other — Estimation only; Median = 7.3, 95% CI 2-sided [2.2 to 13.0] — The Kaplan Meier method was used to estimate the median PFS(in months) for the population. The Greenwood method was used to estimate the confidence limits of the median progression free survival

4. Secondary Outcome: Overall Survival
Description: OS is defined as the duration of time from enrollment to the date of death from any cause. Subjects who were alive or lost to follow-up at the time of the analysis were censored at the last known date they were alive.
Time Frame: From date of treatment start to date of death, or censored as described above; assessed for approximately 3 years
Population: Efficacy analyses were conducted on the population of subjects who began Carboplatin + Abraxane treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin + Abraxane
Number analyzed (Participants) | 11
months | 30 [2.2 to NA] — Upper limit of the confidence interval is not reached due to censoring rate.
Statistical Analysis 1: Comparison: Carboplatin + Abraxane; Test type: Other — Estimation only; Median = 30.0, 95% CI 2-sided [lower limit 2.2] (Upper limit of the confidence interval is not reached due to censoring rate.) — The Kaplan Meier method was used to estimate median OS(in months). The Greenwood method was used to estimate confidence limits of median overall survival

5. Secondary Outcome: Duration of Response
Description: For subjects who achieve a CR or PR, response duration will be measured from the first day of the response until the day on which progressive disease (PD) or death occurred. The censoring method will be the same as that described for PFS.
Time Frame: From date of response to date of progression/death, or censored as described above; assessed for approximately 3 years.
Population: Efficacy analyses were conducted on the population of subjects who began Carboplatin + Abraxane treatment. Duration of response was conducted specifically on those subjects in the efficacy population who achieved objective response (PR or CR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin + Abraxane
Number analyzed (Participants) | 4
months | 10.8 [4.9 to 11.9]
Statistical Analysis 1: Comparison: Carboplatin + Abraxane; Test type: Other — Estimation only; Median = 10.8, 95% CI 2-sided [4.9 to 11.9] — The Kaplan Meier method was used to estimate median duration of response (in months). The Greenwood method was used to estimate confidence limits of median duration of response

6. Secondary Outcome: Duration of Disease Control
Description: For subjects who achieve SD or better, duration of disease control will be measured from the treatment start date until the day on which progressive disease (PD) or death occurred. The censoring method will be the same as that described for PFS.
Time Frame: From date of treatment start to date of progression, or censored as described above; assessed for approximately 3 years
Population: Efficacy analyses were conducted on the population of subjects who began Carboplatin + Abraxane treatment. Duration of disease control was conducted specifically on those subjects in the efficacy population who achieved disease control (stable disease or better).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin + Abraxane
Number analyzed (Participants) | 9
months | 7.3 [3.0 to 13.0]
Statistical Analysis 1: Comparison: Carboplatin + Abraxane; Test type: Other — Estimation only; Median = 7.3, 95% CI 2-sided [3.0 to 13.0] — The Kaplan Meier method was used to estimate median duration of disease control (in months). The Greenwood method was used to estimate confidence limits of median disease control duration

ADVERSE EVENTS:
Time Frame: Baseline, during treatment (up to a planned 18 weeks), and 30 days after last dose of treatment administration
Arm/Group | Carboplatin + Abraxane
All-Cause Mortality (participants affected / at risk) | 6/11
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin + Abraxane (N=11)
Blood bilirubin increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Sepsis (Infections and infestations) | 1
White blood cell decreased (Investigations) | 1
Lung infection (Infections and infestations) | 1
Confusion (Psychiatric disorders) | 1
Fatigue (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin + Abraxane (N=11)
Anemia (Blood and lymphatic system disorders) | 10
Fatigue (General disorders) | 9
Platelet count decreased (Investigations) | 8
Peripheral sensory neuropathy (Nervous system disorders) | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Neutrophil count decreased (Investigations) | 6
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 4
Edema limbs (General disorders) | 4
Diarrhea (Gastrointestinal disorders) | 4
Mucositis oral (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 3
Alkaline phosphatase increased (Investigations) | 3
Weight loss (Investigations) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dizziness (Nervous system disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hypotension (Vascular disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
White blood cell decreased (Investigations) | 2
Bruising (Injury, poisoning and procedural complications) | 2
Skin infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Lung infection (Infections and infestations) | 2
Chills (General disorders) | 2
Localized edema (General disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Sinus tachycardia (Cardiac disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Blood bilirubin increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Gum infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Mucosal infection (Infections and infestations) | 1
Fever (General disorders) | 1
Infusion related reaction (General disorders) | 1
Neck edema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 — oral candidiasis
Oral hemorrhage (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Conjunctivitis (Eye disorders) | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Confusion (Psychiatric disorders) | 1
Headache (Nervous system disorders) | 1
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neuralgia (Nervous system disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 — Contact dermatitis
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-11-11): https://cdn.clinicaltrials.gov/large-docs/05/NCT02328105/Prot_SAP_000.pdf
  • Informed Consent Form (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT02328105/ICF_001.pdf